CLINICAL TRIAL: NCT03124147
Title: Optimizing Transcranial Direct Current Stimulation for Motor Recovery From Severe Post-stroke Hemiparesis
Brief Title: Optimizing Transcranial Direct Current Stimulation for Motor Recovery From Hemiparesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumy Sawaki (Other)
Responsible Party: Sponsor-Investigator, Lumy Sawaki, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 11CRP7220009
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Stroke; Cerebrovascular Accident
Keywords: motor recovery; neuroplasticity; chronic; human; noninvasive brain stimulation; neuromodulation
MeSH Terms: conditions — Stroke; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Anodal tDCS with motor training (Active Comparator): 20 minutes of anodal transcranial direct current stimulation applied to the ipsilesional hemisphere (intervention) paired with 3 hours of intensive, task-oriented upper extremity motor training. Transcranial direct current stimulation will be delivered using the Neuroconn Eldith stimulator by Magstim.
  Interventions: Device: Neuroconn Eldith stimulator by Magstim
- Cathodal tDCS with motor training (Active Comparator): 20 minutes of cathodal transcranial direct current stimulation applied to the contralesional hemisphere (intervention) paired with 3 hours of intensive, task-oriented upper extremity motor training. Transcranial direct current stimulation will be delivered using the Neuroconn Eldith stimulator by Magstim.
  Interventions: Device: Neuroconn Eldith stimulator by Magstim
- Dual tDCS with motor training (Active Comparator): 20 minutes of anodal transcranial direct current stimulation applied to the ipsilesional hemisphere and cathodal transcranial direct current stimulation applied to the contralesional hemisphere (intervention) paired with 3 hours of intensive, task-oriented upper extremity motor training. Transcranial direct current stimulation will be delivered using the Neuroconn Eldith stimulator by Magstim.
  Interventions: Device: Neuroconn Eldith stimulator by Magstim
- Sham tDCS with motor training (Sham Comparator): 20 minutes of sham transcranial direct current stimulation applied to the ipsilesional hemisphere (intervention) paired with 3 hours of intensive, task-oriented upper extremity motor training. Transcranial direct current stimulation will be delivered using the Neuroconn Eldith stimulator by Magstim.
  Interventions: Device: Neuroconn Eldith stimulator by Magstim

INTERVENTIONS:
Device: Neuroconn Eldith stimulator by Magstim — Transcranial direct current stimulation to the ipsilesional hemisphere, contralesional hemisphere, or both, paired with task-oriented therapy.

SUMMARY:
This study will compare the effectiveness of different polarities of transcranial direct current stimulation paired with intensive motor training in recovery of upper extremity function in individuals with severe post-stroke hemiparesis. The hypothesis is that more severely impaired individuals will derive greater benefit from anodal stimulation of the ipsilesional hemisphere or cathodal stimulation of the contralesional hemisphere than dual stimulation (anodal applied to the ipsilesional hemisphere and cathodal applied to the contralesional hemisphere.)

DETAILED DESCRIPTION:
This study has 2 aims: 1) determine which transcranial direct current stimulation (tDCS) electrode configuration is most effective in combination with motor training to promote motor recovery from severe post-stroke hemiparesis; and 2) begin to clarify the extent to which baseline transcranial magnetic stimulation (TMS) measures predict response to tDCS, as well as the effects of tDCS paired with motor training on TMS measures of motor cortical organization.

To accomplish these aims, the investigators will recruit 36 human subjects with severe post-stroke hemiparesis and assign each subject to 1 of 4 tDCS conditions (anodal excitatory ipsilesional; cathodal inhibitory contralesional; a combination of anodal excitatory ipsilesional during cathodal inhibitory contralesional; or sham). Each subject will undergo a 20-minute stimulation session once a day for 10 days over a 2-week period. Each session will be followed by 3 hours of intensive, task-oriented upper extremity motor training.

Outcome measures for this study include TMS motor cortical maps and standardized tests of motor performance. The investigators hypothesize that all groups will show improvement in all measures; however, both the anodal excitatory ipsilesional group and the cathodal inhibitory contralesional group will show significantly greater improvement compared with the other 2 groups. The investigators will also find evidence clarifying whether the presence or absence of motor-evoked potentials (MEPs) has predictive value regarding which tDCS configuration would be most effective for a particular subject.

ELIGIBILITY:
Inclusion Criteria:

* Chronic stroke patients
* Single stroke
* Chronic (more than 12 months after from stroke)
* At least 18 years old, but there is no upper age range for this project.
* Participants NOT able to extend the affected metacarpophalangeal joints at least 10° and the wrist 20°.

Exclusion Criteria:

* History of head injury with loss of consciousness, seizure, severe alcohol or drug abuse, psychiatric illness
* Within 3 months of recruitment, use of drugs known to exert detrimental effects on motor recovery
* Cognitive deficit severe enough to preclude informed consent
* Positive pregnancy test or being of childbearing age and not using appropriate contraception
* Participants with history of untreated depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change in Fugl Meyer Assessment | Score change after 10 days of intervention compared to baseline; Score change after 1-month after the intervention compared to baseline

SECONDARY OUTCOMES:
Change in Action Research Arm Test | Score change after 10 days of intervention compared to baseline; Score change after 1-month after the intervention compared to baseline
Change in Stroke Impact Scale | Score change after 10 days of intervention compared to baseline; Score change after 1-month after the intervention compared to baseline

IPD SHARING:
Plan to Share IPD: No